CLINICAL TRIAL: NCT00839436
Title: Interleukin-7 (CYT107) Treatment of Idiopathic CD4 Lymphocytopenia: Expansion of CD4 T Cells (ICICLE)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Bankruptcy of Drug manufacturer: Drug not available
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090069; 09-I-0069
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Results first posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Idiopathic CD4+ T-Lymphocytopenia
Keywords: Idiopathic CD4+ T-Lymphocytopenia; Interleukin-7; Clinical Trial; T-Lymphocytes; Idiopathic CD4 Lymphocytopenia (ICL); ICL
MeSH Terms: conditions — T-Lymphocytopenia, Idiopathic CD4-Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 3 microgram/kg CYT107 (Experimental): 3 microgram/kg CYT107
  Interventions: Drug: CYT107
- 10 microgram/kg CYT107 (Experimental): 10 microgram/kg CYT107
  Interventions: Drug: CYT107
- 20 microgram/kg CYT107 (Experimental): 20 microgram/kg CYT107
  Interventions: Drug: CYT107

INTERVENTIONS:
Drug: CYT107

SUMMARY:
Background:

* Idiopathic CD4 lymphocytopenia (ICL) is a condition in which patients have low levels of T cells, a type of white blood cell that helps fight infection. Animal studies have shown that an experimental drug Interleukin 7 (IL-7), which is named CYT107, can increase the number and function of T cells. CYT107, however, has not been used in people with ICL.

Objectives:

* To determine the safety of CYT107 in people with ICL.
* To determine whether CYT107 will increase the number and function of T cells in people with ICL.

Eligibility:

* Patients 18 years of age and older diagnosed with ICL and who are at risk of becoming sick because of this condition are eligible for this study. In addition, patients must not be pregnant, or have other illnesses that would cause low CD4 T cell counts, such as human immunodeficiency virus (HIV) or human T-lymphotrophic virus (HTLV) infection.

Design:

* The initial screening visit will include the following examinations and tests:
* A complete physical exam and medical history
* Blood analysis, including CD4 T cell count; complete blood count and additional blood tests to determine clotting ability and blood composition; thyroid, liver, kidney, and pancreatic function tests; HIV and HTLV tests; and tests for anti-IL-7 antibodies that block normal IL-7 activity
* Routine urine test
* Urine or blood pregnancy test for women
* Chest X-ray
* Electrocardiogram
* Spleen ultrasound.
* The baseline visit will include blood tests to determine levels of each of the major types of antibodies, a test of genetic background, and more detailed CD4 and protein analysis. In addition, leukapheresis (a procedure to collect large numbers of immune cells without red blood cells) will be done. Participants will also have the option of having colon and lymph node biopsies.
* The schedule will be as follows:
* Weeks 1, 2, and 3 (Cycle 1): Three weekly IL-7 dosing visits.
* Weeks 5, 8, and 12: Follow-up visits.
* Weeks 24, 25, and 26 (Cycle 2): Three more weekly IL-7 dosing visits.
* Weeks 28, 31, and 35: Follow-up visits.
* Week 48: End of study visit.
* Tests conducted before getting IL-7 will be repeated during the IL-7 cycles and follow-up visits to compare with earlier values. Optional colon and lymph node biopsies done at baseline will be repeated 1 6 weeks prior to Cycle 2 and 1 6 weeks prior to Week 48.

DETAILED DESCRIPTION:
Interleukin-7 (CYT107) Treatment of Idiopathic CD4 Lymphocytopenia: Expansion of CD4 T Cells (ICICLE) is a Phase I/IIa open-label, single arm clinical trial evaluating the safety profile of glycosylated recombinant human interleukin-7 (rhIL-7) as an immunostimulatory therapy in patients with idiopathic CD4 T cell lymphocytopenia (ICL) at risk of disease progression. Secondary analyses will assess the immunostimulatory effects of rhIL-7 on T cell number and function.

ICL was first characterized in the early 1990 s and is a primary immune disorder of CD4 T cell lymphocytopenia (less than 300 cells/microL or less than 20% of lymphocytes), which is not due to any known infectious process, exogenous medication, autoimmune cytopenia, or other underlying disorder associated with lymphocytopenia. ICL patients are at risk for a wide spectrum of opportunistic and other serious infections, autoimmune disorders, and other types of lymphocytopenia. At present, no validated treatment exists for ICL, and treatment is directed primarily toward infectious complications once they arise. A first-generation form of rhIL-7 was shown in pre-clinical and Phase I studies in oncology and human immunodeficiency virus (HIV)-infected patients to be well tolerated in repeated dose trials, with long-lasting increases in both CD4 and CD8 T cells. CYT107 is a second-generation rhIL-7 product made by Cytheris via a recombinant mammalian cell culture system.

DESIGN - Open-label, single-arm, Phase I/IIa interventional clinical trial. Participants will be evaluated at baseline (prior to study treatment) and according to the protocol follow-up schedule, receiving a total of 2 cycles of rhIL-7 (CYT107) during the induction phase and up to 8 cycles during the maintenance phase. Safety assessments of rhIL-7 will be the primary focus at each study visit, with secondary analyses of immune parameters, including changes from baseline in T cell number and function at Weeks 24 and 48.

DURATION - Enrollment is expected to take 3 to 4 years. Each volunteer will be followed for at least 48 weeks. Thus, total duration of the study will be approximately 5 years.

SAMPLE SIZE - Approximately 35-40 patients will be screened over a 3-year period to achieve the desired sample of 18 ICL patients, allowing for a primary safety assessment of CYT107 in this Phase I/IIa clinical trial, as well as exploring the immunomodulatory effects of rhIL-7.

POPULATION - Men and women, aged greater than or equal to 18 years, with a confirmed diagnosis of ICL (CD4 less than 300 cells/micromL or less than 20% of lymphocytes) deemed at risk for complications due to concurrent CD8 T cell lymphocytopenia and/or history of opportunistic or otherwise serious infection, without autoimmunity or hematologic or lymphoid malignancy.

REGIMEN - During the induction phase, subjects will receive 2 cycles of subcutaneous rhIL-7 dosed once weekly for 3 weeks in a dose escalation fashion: 3 microg/kg (first 3 subjects-completed), 10 microg/kg (next 5 subjects-completed) and 20 microg/kg (last 5 subjects), with an additional 5 subjects at the highest achieved dose level. Cycles of rhIL-7 will be administered starting at Week 1 and Week 24.

For subjects who tolerate the induction phase and elect to participate in the

maintenance phase, additional cycles of rhIL-7 may be offered at 3-6 month

intervals. These participants will receive rhIL-7 at the highest dose for which at

least 8 weeks of safety data for 5 subjects has been reviewed provided no more

than 1 DLT is reported.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Age greater than or equal to 18 years
2. CD4 T cell count less than 300 cells/microL or less than 20% of total T lymphocytes on 2 occasions at least 6 weeks apart (and at the time of screening) in the absence of any illness accounting for CD4 lymphocytopenia
3. ICL diagnosis that indicates a risk for disease progression, defined as one or both of the following:

   * CD8 T cell lymphocytopenia (less than 180 cells/microL)
   * History of opportunistic or otherwise significant infection (e.g., AIDS-defining or highly morbid illnesses, such as Cryptococcus or Mycobacteria infection, severe herpes zoster, JC virus causing progressive multifocal leukoencephalopathy, Kaposi s sarcoma, or severe human papilloma virus condylomata)
4. HIV-1 and HIV-2 seronegativity and below detection of HIV-1 viral load
5. HTLV-1 and HTLV-2 seronegativity
6. Adequate venous access, as determined by the study team, although participants unable to undergo leukapheresis will not be excluded
7. Normal thyroid-stimulating hormone (TSH)
8. Negative serum or urine pregnancy test at time of study enrollment for women of childbearing potential
9. Ability to understand and give informed consent
10. Capacity and willingness to adhere to study procedures, including scheduled follow-up visits
11. Willingness to allow blood and tissue sample storage
12. Established primary care provider

EXCLUSION CRITERIA:

1. History of prior cytotoxic, chemotherapeutic, immunosuppressant (e.g., systemic corticosteroids), immunomodulatory (e.g., IL-2, IL-7, interferon-gama), or growth factor therapy within the last 6 months; chemotherapy or immunomodulatory therapy given to treat an underlying disease or condition may be permitted at the protocol team's discretion, provided diagnosis of ICL was established prior to starting this treatment. The treatment has been stable for over 6 months and is being administered at stable doses as maintenance therapy.
2. History of prior participation in another investigational intervention study within the last 6 months. Co-enrollment in other NIAID stem cell mobilization protocols will be permitted at the protocol team s discretion, but CYT107 may be dosed no sooner than 6 months after last dose of that protocol s medications have been given.
3. Active uncontrolled opportunistic infection at the time of enrollment
4. Current or recent history (less than 28 days prior to screening) of a viral, bacterial, parasitic or fungal infection requiring hospitalization and/or systemic treatment, other than long-term maintenance pharmacotherapy
5. Serious illness requiring systemic treatment and/or hospitalization within 56 days (8 weeks) of screening, unless the subject is clinically stable, in the opinion of the Principal Investigator, and has completed therapy or has been on appropriate therapy for greater than 28 days (4 weeks) prior to screening
6. Current or history of hematologic or lymphoid (lymphoma) malignancy
7. Established or planned pregnancies or refusal to use effective birth control (e.g., barrier methods, oral contraceptives, intrauterine devices) for the duration of study involvement, regardless of gender
8. Concurrent breastfeeding
9. Renal insufficiency (e.g., estimated glomerular filtration rate less than 60 mL/min/1.73 m(2))
10. Any of the following screening laboratory abnormalities: platelets less than 100,000 cells/microL; lipase greater than 1.5 times the ULN; AST, ALT, or alkaline phosphatase greater than 2.5 times the ULN; total bilirubin greater than 1.5 times the ULN
11. History of splenectomy or hematologic disease associated with hypersplenism, such as alpha- or beta-thalassemia, hereditary spherocytosis, Gaucher s disease, or autoimmune hemolytic anemia
12. Cirrhosis of any origin, including alcoholic or non-alcoholic steatohepatitis, either suspected by history or histologically proven
13. History of hepatitis B or C infection, i.e., positive hepatitis B surface antigen, positive anti-hepatitis B core antibody with a detectable hepatitis B DNA viral load, positive anti-hepatitis C antibody and/or detectable hepatitis C RNA viral load (subjects who became negative for hepatitis B DNA or hepatitis C RNA following anti-viral treatment will not qualify for study treatment)
14. Need for anticoagulant medication (e.g., warfarin, heparin), other than aspirin, clopidogrel, or other antiplatelet agent as CYT107 may co-precipitate with heparin if taken together.
15. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements (subjects must agree to refrain from substance abuse use during the entire course of the study)
16. Past or current psychiatric illness that, in the opinion of the investigator, would interfere with protocol adherence or the ability and willingness to give written informed consent
17. Current autoimmune conditions requiring systemic (oral, injection, or other parenteral) therapy, as well as psoriasis and optic neuritis regardless of treatment and/or a diagnosis of systemic lupus erythematous based on the screening rheumatologic work up.
18. Cardiac, pulmonary, thyroid, renal, hepatic, neurological (central or peripheral) disease or disorder of hemostasis requiring therapy and considered to be significant by the protocol team
19. History of cardiovascular disease, arrhythmias, or clinically significant ECG abnormalities, including a corrected QT interval (QTc) greater than or equal to 470 milliseconds
20. Family history consistent with an inherited cardiomyopathy or arrhythmia such as the following:

    * Arrhythmogenic Right Ventricular Dysplasia (ARVD)
    * Brugada syndrome (BrS)
    * Congenital Long QT (LQT)
    * Congenital Short QT intervals (SQT)
    * Early Repolarization Syndrome
    * Idiopathic Ventricular Fibrillation (IVF)
21. Uncontrolled hypertension (i.e., resting systolic blood pressure greater than160 mmHg or resting diastolic blood pressure greater than 90 mmHg), despite pharmacologic antihypertensive treatment, confirmed with a second blood pressure measurement done later in the same day.
22. Evidence of circulating neutralizing anti-IL-7 antibodies (prior to initial rhIL-7 administration)

To be eligible for rhIL-7 administration, all Exclusion Criteria are prohibited. However, for the purpose of performing baseine pre-IL-7 procedures certain Exclusion Criteria designed to minimize specific complications from rhIL-7 (e.g., autoimmune or lymphoproliferative complications) but that do not increase the risk associated with these procedures are permitted, as baseline procedures will be done prior to IL-7 administration: #6, #11, through #13, #17, #18, #20, #22.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-02; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia M Sheikh, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Smith DK, Neal JJ, Holmberg SD. Unexplained opportunistic infections and CD4+ T-lymphocytopenia without HIV infection. An investigation of cases in the United States. The Centers for Disease Control Idiopathic CD4+ T-lymphocytopenia Task Force. N Engl J Med. 1993 Feb 11;328(6):373-9. doi: 10.1056/NEJM199302113280601. PMID 8093633
- [Background] Walker UA, Warnatz K. Idiopathic CD4 lymphocytopenia. Curr Opin Rheumatol. 2006 Jul;18(4):389-95. doi: 10.1097/01.bor.0000231908.57913.2f. PMID 16763460
- [Background] Bofill M, Janossy G, Lee CA, MacDonald-Burns D, Phillips AN, Sabin C, Timms A, Johnson MA, Kernoff PB. Laboratory control values for CD4 and CD8 T lymphocytes. Implications for HIV-1 diagnosis. Clin Exp Immunol. 1992 May;88(2):243-52. doi: 10.1111/j.1365-2249.1992.tb03068.x. PMID 1349272
- [Derived] Sheikh V, Porter BO, DerSimonian R, Kovacs SB, Thompson WL, Perez-Diez A, Freeman AF, Roby G, Mican J, Pau A, Rupert A, Adelsberger J, Higgins J, Bourgeois JS Jr, Jensen SM, Morcock DR, Burbelo PD, Osnos L, Maric I, Natarajan V, Croughs T, Yao MD, Estes JD, Sereti I. Administration of interleukin-7 increases CD4 T cells in idiopathic CD4 lymphocytopenia. Blood. 2016 Feb 25;127(8):977-88. doi: 10.1182/blood-2015-05-645077. Epub 2015 Dec 16. PMID 26675348

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3 mcg/kg Cohort | 10 mcg/kg Cohort | 20 mcg/kg Cohort
Started | 3 | 5 | 1
Completed | 2 | 4 | 0
Not Completed | 1 | 1 | 1
Not completed — Developed exclusionary condition | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Study drug no longer available | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 mcg/kg Cohort | 10 mcg/kg Cohort | 20 mcg/kg Cohort | Total
Number analyzed (Participants) | 3 | 5 | 1 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 1 | 8
  >=65 years | 0 | 1 | 0 | 1
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49 [23 to 51] | 56 [44.5 to 63.5] | 33 [33 to 33] | 51 [33.5 to 56.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 7
  Male | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 1 | 9
CD4 T cell count [Median (Inter-Quartile Range); unit: cells/microliter] | 13 [10 to 18] | 52 [20 to 183.5] | 15 [15 to 15] | 18 [14 to 116]

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events and Toxicities Associated With CYT107.
Time Frame: 48 weeks per patient with a 3-4 year enrollment period
Measure: Number; unit: Events
Arm/Group | 3 mcg/kg Cohort | 10 mcg/kg Cohort | 20 mcg/kg Cohort
Number analyzed (Participants) | 3 | 5 | 1
Events
  Grade 5 Adverse Events | 0 | 0 | 0
  Grade 4 Adverse Events | 0 | 0 | 0
  Grade 3 Adverse Events | 3 | 0 | 0
  Grade 2 Adverse Events | 21 | 45 | 0
  Grade 1 Adverse Events | 103 | 112 | 8

2. Other Pre Specified Outcome: Change: CD4/CD8 T Cell Cts After CYT107; in Immunophenotype (Naive, Memory, Regulatory T Cell Subsets) & Amp; Antigen-specific T Cell Function After CYT107; in T Cell Activation/Proliferation Status & Amp; TCR Repertoire After CYT107; ...
Time Frame: 48 weeks per patient with a 3-4 year enrollment period
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | 3 mcg/kg Cohort | 10 mcg/kg Cohort | 20 mcg/kg Cohort
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/5 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mcg/kg Cohort (N=3) | 10 mcg/kg Cohort (N=5) | 20 mcg/kg Cohort (N=1)
Systemic Lupus Erythematosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute hypersensitivity reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mcg/kg Cohort (N=3) | 10 mcg/kg Cohort (N=5) | 20 mcg/kg Cohort (N=1)
lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 2 (8) | 2 (2) | 1 (1)
lymphadenopathy (Blood and lymphatic system disorders) | 2 (5) | 1 (3) | 1 (1)
pyrexia (General disorders) | 0 (0) | 1 (3) | 1 (1)
injection site reaction (General disorders) | 3 (6) | 5 (20) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (2)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
hyperhydrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 2 (2) | 1 (1) | 0 (0)
injection site recall reaction (General disorders) | 2 (5) | 1 (1) | 0 (0)
Blood bicarbonate abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
panic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
pain (General disorders) | 1 (1) | 2 (2) | 0 (0)
hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (2) | 0 (0)
angina pectoris (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
tooth disorder (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0)
tenderness (General disorders) | 1 (1) | 3 (4) | 0 (0)
palpitations (Cardiac disorders) | 0 (0) | 2 (4) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 3 (6) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (6) | 0 (0)
nausea (Gastrointestinal disorders) | 2 (2) | 2 (6) | 0 (0)
haemoglobin decreased (Investigations) | 3 (13) | 2 (7) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (7) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (8) | 0 (0)
fatigue (General disorders) | 2 (4) | 3 (8) | 0 (0)
injection site pruritis (General disorders) | 0 (0) | 4 (12) | 0 (0)
acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
alveolar osteitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
anogenital dysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
apthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Breast discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
dry moutn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
external ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
hypocalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
libido increased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
pyuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
supplementation therapy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
eye disorder (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
hot flush (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
hypoglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
proteinuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes